CLINICAL TRIAL: NCT04230538
Title: A Prospective Randomised Control Study in 6-16 Year Old Children Presenting to Sheffield Children's NHSFT With Stable Ankle Injuries That Would Otherwise Have Received Cast Immobilisation.
Brief Title: Plaster Cast Versus DJO Walker in Paediatric Ankle Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCH/12/070
Record Dates: First submitted 2015-04-23; First posted 2020-01-18 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Ankle Sprain Strain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DJO Walker (Experimental): Application of DJO Walker
  Interventions: Device: DJO Walker
- Traditional plaster cast (Active Comparator): Application of traditional plaster cast
  Interventions: Device: Traditional plaster cast

INTERVENTIONS:
Device: DJO Walker
  Arms: DJO Walker
Device: Traditional plaster cast
  Arms: Traditional plaster cast

SUMMARY:
Present treatment of children with stable ankle and foot injuries very often involves a period in plaster cast(s). In the last decade in adult patients this has been superceded in many instances by the use of a removable foot brace/splint.

There are many benefits to this approach including progressive rehabilitation, reduced costs in materials and personnel, improved hygiene and adaptability of fit. The use of such a splint has not been investigated in children and this project aims to assess the value of introducing this as a treatment mode through the analysis of outcomes between traditional cast treatment and the newer removable brace/splint treatment. The outcomes will include patients' preferences, clinical results and relative costings.

DETAILED DESCRIPTION:
The study is a longitudinal cohort study of all eligible ankle injuries per the eligibility criteria presenting to Sheffield Children's NHS Fountain Trust. These children and their parents/carers are presented with an information sheet regarding the study and are then invited to enter the study.

Once consented - by appropriately trained research and/or clinical staff - those recruited are treated in either cast or boot on the basis of block randomisation.

Patients are followed up per protocol and outcomes completed by patients and clinicians.

Study information is kept securely for future analysis and write up.

ELIGIBILITY:
Inclusion Criteria:

1. 6-16 years
2. foot size has to be large enough for the smallest available DJO Walker
3. presentation to the Sheffield Children's Hospital Emergency Department or Fracture Clinic (some patients present directly to the fracture clinic if they have been injured elsewhere (eg. on holiday or in competitions)
4. acute injuries (less than 72 hours old)
5. stable ankle injuries. This is all ankle sprains and all stable undisplaced ankle fractures. The key here is that the patient would be able to weightbear in cast/DJO Walker without detriment to the ankle injury, pain permitting
6. signed consent

Exclusion Criteria:

1. <6 and >16
2. foot size too small for DJO Walker
3. any unstable ankle injury
4. any ankle injury that could not be treated weightbearing in cast/aircast boot (pain permitting)
5. patients/carers unwilling to participate in the study

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-03-12 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
To compare the plaster cast intervention versus the DJO Walker intervention | 3 months
  Patient and Carer Treatment Evaluation Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mark Flowers, Principal Investigator — Investigator
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, Sheffield (South Yorkshire District), United Kingdom